CLINICAL TRIAL: NCT03868241
Title: Randomized Controlled Open-label Trial Assessing the Efficacy of a Bundle of Coated Devices to Reduce Nosocomial Infections in the Intensive Care Unit
Brief Title: Coated Devices to Decrease Infection in the Intensive Care Unit
Acronym: CRITIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Bactiguard AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRITIC_PILOT
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Critically Ill
Keywords: sepsis; ventilator-associated pneumonia; catheter related bloodstream infection; urinary catheter-related infection
MeSH Terms: conditions — Critical Illness; Sepsis; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bactiguard-coated Devices (Experimental): Patients will receive endotracheal tube, central venous catheter and urinary cather coated with gold, silver and palladium (Bactiguard coating)
  Interventions: Device: Coated devices
- Control (Placebo Comparator): Shelf endotracheal tube, central venous catheter and urinary cather available at each intensive care unit without any type of coating designed to prevent infection
  Interventions: Device: Control

INTERVENTIONS:
Device: Coated devices — Gold-silver-palladium coated devices (endotracheal tube, central venous catheter and urinary catheter) will be used whenever necessary. All three devices are required to be inserted as soon as possible after randomization and need for all three devices are the main inclusion criteria
  Arms: Bactiguard-coated Devices
Device: Control — Devices without coating available at each participating intensive care unit
  Arms: Control

SUMMARY:
Pilot explanatory, randomized, open label, controlled trial. Critically ill patients which will demand placement of invasive devices for organ support (endotracheal tube, central venous catheter and urinary Foley catheter) will be randomized 1:1 to receive coated (Bactiguard®) or habitual (non-coated) devices.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the intensive care unit which will require simultaneous insertion of all three devices (endotracheal tube, central venous catheter and urinary catheter) due to illness severity as defined by the attending physician.

Exclusion Criteria:

* Patients admitted to the intensive care unit for more than 48 hours or admitted in the hospital for more than seven days
* Presence of any of the invasive devices (endotracheal tube, central venous catheter or urinary catheters) before randomization and absence of the intention to exchange the devices;
* Previous use of any type of coated devices;
* Age < 18 years;
* Known pregnancy
* Known allergy to gold, silver and palladium;
* Suspected or confirmed brain death;
* Previously enrolled in the study

Newly added exclusion criteria in version 2.0:

* Severe chronic pulmonary obstructive disease which may limit catheter site selection
* Previous irradiation and/or thrombosis in site selected for catheter insertion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants recruited in each center during the trial | Through study completion, an average of 1 year
  Assess the recruitment rate
Number of participants admitted to the intensive care unit that requires simultaneous insertion of endotracheal tube, central venous catheter and urinary catheter | Through study completion, an average of 1 year
  Assess how many patients admitted to the intensive care unit will demand insertion of endotracheal tube, urinary catheter and central venous catheter after admission in all patients
Feasibility - Occurence of sepsis | 28 days
  Occurrence of sepsis after admission in patients that require all three devices to be inserted in all patients

SECONDARY OUTCOMES:
Sepsis | 28 days
  Occurrence of sepsis after randomization (defined as infection plus organ failure)
Occurence of ventilator-associated pneumonia | 28 days
  Occurence of ventilator-associated pneumonia by radiographic and clinical criteria
Occurence of central venous catheter-related bloodstream infection | 28 days
  Occurence of central venous catheter-related bloodstream infection using Brazilian regulatory agency criteria
Occurence of urinary catheter-related infection | 28 days
  Occurence of urinary catheter-related infection defined as positive urinary culture coupled with fever and without any other infection source
Rate of composite endpoint of ventilator-associated pneumonia and/or central venous catheter-related bloodstream infection and/or urinary catheter-related infection | 28 days
  Occurrence of any of the infections above
Antibiotic-free days | 28 days
  Number of days not receiving antibiotics
Number of patients that die in Intensive Care Unit | Through intensive care unit stay, an average of 28 days
  Mortality during intensive care unit stay
Number of patients that die during hospital stay | Through hospital stay, an average of 40 days
  Mortality during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Biasi, MD/PhD, Study Director — Hospital do Coração
Locations (6):
- Brazil (6):
  - Hospital de Base de São José do Rio Preto, Rio Preto, São Paulo
  - Hospital do Coração, São Paulo, São Paulo
  - AC Camargo Câncer Center, São Paulo
  - Hospital da Luz, São Paulo
  - Hospital Paulistano, São Paulo
  - Hospital São Paulo - UNIFESP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zampieri FG, de Oliveira NE, Nassar AP Jr, de Oliveira Manoel AL, Grion C, Lacerda FH, Maia I, Thompson M, Giancursi TS, de Aquino Martins P, Lisboa T, Abait T, Damiani LP, Machado FR, Cavalcanti AB; BRICNet. Bundle of Coated Devices to Reduce Nosocomial Infections in the Intensive Care Unit. CRITIC Pilot Randomized Controlled Trial. Ann Am Thorac Soc. 2020 Oct;17(10):1257-1263. doi: 10.1513/AnnalsATS.202003-206OC. PMID 32526149

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03868241/SAP_000.pdf